CLINICAL TRIAL: NCT04432207
Title: An Open Label, Multi-Center, Dose Escalation/Expansion, Phase 1/1b Study of IMU-201, a B-Cell Immunotherapy As Monotherapy or in Combination with Atezolizumab with or Without Chemotherapy, in Adults with Non- Small Cell Lung Cancer (IMPrinter)
Brief Title: A Study of IMU-201 (PD1-Vaxx), a B-Cell Immunotherapy, in Adults with Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imugene Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMU.201.101
Record Dates: First submitted 2020-05-10; First posted 2020-06-16 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-01

CONDITIONS: Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Stage IIIB; Non-small Cell Lung Cancer Stage IV; Squamous Non-small-cell Lung Cancer; Large Cell Carcinoma Lung; Adenocarcinoma Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (13):
- Dose Escalation: Monotherapy Cohort 1 (Experimental): 10 μg/dose IMU-201 as a 0.5 mL PD1-Vaxx injection Progressed on/after ICI, TPS/TC ≥50% or IC ≥10%
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 1
- Dose Escalation: Monotherapy Cohort 2 (Experimental): 50 μg/dose IMU-201 as a 0.5 mL PD1-Vaxx injection Progressed on/after ICI, TPS/TC ≥50% or IC ≥10%
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 1
- Dose Escalation: Monotherapy Cohort 3 (Experimental): 100 μg/dose IMU-201 as a 0.5 mL PD1-Vaxx injection Progressed on/after ICI, TPS/TC ≥50% or IC ≥10%
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 1
- Dose Expansion Monotherapy (Experimental): mOBD (TBD) dose IMU-201 as a 0.5 mL PD1-Vaxx injection Progressed on/after ICI, TPS/TC ≥50% or IC ≥10%
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 1
- Dose Escalation Arm 1: Combination with atezolizumab Cohort 1 (Experimental): 10 μg/dose IMU-201 as a 0.5 mL PD1-Vaxx injection with atezolizumab 840 mg Naïve to ICI or Progressed on/after ICI, TPS/TC ≥50% or IC ≥10%
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 2; Drug: Atezolizumab
- Dose Escalation Arm 1: Combination with atezolizumab Cohort 2 (Experimental): 50 μg/dose IMU-201 as a 0.5 mL PD1-Vaxx injection with atezolizumab 840 mg Naïve to ICI or Progressed on/after ICI, TPS/TC ≥50% or IC ≥10%
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 2; Drug: Atezolizumab
- Dose Escalation Arm 1: Combination with atezolizumab Cohort 3 (Experimental): Cohort 3: 100 μg/dose IMU-201 as a 0.5 mL PD1-Vaxx injection with atezolizumab 840 mg Naïve to ICI or Progressed on/after ICI, TPS/TC ≥50% or IC ≥10%
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 2; Drug: Atezolizumab
- Dose Escalation Arm 2: Combination with atezolizumab and chemotherapy Cohort 1 (Experimental): 10 μg/dose IMU-201 as a 0.5 mL PD1-Vaxx injection with atezolizumab 840 mg and SOC chemotherapy Naïve to ICI, Any PD-L1 Level
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 3; Drug: Atezolizumab; Drug: Standard of care chemotherapy
- Dose Escalation Arm 2: Combination with atezolizumab and chemotherapy Cohort 2 (Experimental): 50 μg/dose IMU-201 as a 0.5 mL PD1-Vaxx injection with atezolizumab 840 mg and SOC chemotherapy Naïve to ICI, Any PD-L1 Level
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 3; Drug: Atezolizumab; Drug: Standard of care chemotherapy
- Dose Escalation Arm 2: Combination with atezolizumab and chemotherapy Cohort 3 (Experimental): 100 μg/dose IMU-201 as a 0.5 mL PD1-Vaxx injection with atezolizumab 840 mg and SOC chemotherapy Naïve to ICI, Any PD-L1 Level
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 3; Drug: Atezolizumab; Drug: Standard of care chemotherapy
- Dose Expansion Arm 1: Combination with atezolizumab (Experimental): cOBD (TBD) dose IMU-201 as a 0.5 mL PD1-Vaxx injection with atezolizumab 840 mg Progressed on/after ICI, TPS/TC ≥50% or IC ≥10%
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 2; Drug: Atezolizumab
- Dose Expansion Arm 2: Combination with atezolizumab (Experimental): cOBD (TBD) dose IMU-201 as a 0.5 mL PD1-Vaxx injection with atezolizumab 840 mg Naïve to ICI, TPS/TC ≥50% or IC ≥10%
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 2; Drug: Atezolizumab
- Dose Expansion Arm 3: Combination with atezolizumab and chemotherapy (Experimental): cOBD (TBD) dose IMU-201 as a 05 mL PD1-Vaxx injection with atezolizumab 840 mg and SOC chemotherapy Naïve to ICI, Any PD-L1 Level
  Interventions: Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 3; Drug: Atezolizumab; Drug: Standard of care chemotherapy

INTERVENTIONS:
Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 1 — IMU-201 consists of APi2568 (lyophilized IMU-201) dissolved in WFI and emulsified with the adjuvant (Montanide ISA 720 VG) to produce PD1-Vaxx. IMU-201 will be administered as PD1-Vaxx intramuscularly into the deltoid region of the upper arm on Days 1, 15, 29, 64 and thereafter every 63 days until discontinuation from study.
  Other Names: PD1-Vaxx; APi2568
  Arms: Dose Escalation: Monotherapy Cohort 1; Dose Escalation: Monotherapy Cohort 2; Dose Escalation: Monotherapy Cohort 3; Dose Expansion Monotherapy
Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 2 — IMU-201 consists of APi2568 (lyophilized IMU-201) dissolved in WFI and emulsified with the adjuvant (Montanide ISA 720 VG) to produce PD1-Vaxx. IMU-201 will be administered as PD1-Vaxx intramuscularly into the deltoid region of the upper arm on Days 1, 15, 29, 57 and thereafter every subsequent 63 days until discontinuation from study.
  Other Names: PD1-Vaxx; APi2568
  Arms: Dose Escalation Arm 1: Combination with atezolizumab Cohort 1; Dose Escalation Arm 1: Combination with atezolizumab Cohort 2; Dose Escalation Arm 1: Combination with atezolizumab Cohort 3; Dose Expansion Arm 1: Combination with atezolizumab; Dose Expansion Arm 2: Combination with atezolizumab
Biological: IMU-201 (administered as PD1-Vaxx) - Regimen 3 — IMU-201 consists of APi2568 (lyophilized IMU-201) dissolved in WFI and emulsified with the adjuvant (Montanide ISA 720 VG) to produce PD1-Vaxx. IMU-201 will be administered as PD1-Vaxx intramuscularly into the deltoid region of the upper arm on Days 1, 15, 29, 57 and thereafter every 56 or 63 days until discontinuation from study.
  Other Names: PD1-Vaxx; APi2568
  Arms: Dose Escalation Arm 2: Combination with atezolizumab and chemotherapy Cohort 1; Dose Escalation Arm 2: Combination with atezolizumab and chemotherapy Cohort 2; Dose Escalation Arm 2: Combination with atezolizumab and chemotherapy Cohort 3; Dose Expansion Arm 3: Combination with atezolizumab and chemotherapy
Drug: Atezolizumab — Atezolizumab will be administered every 2 weeks (Q2W) starting Day 15 until discontinuation from study.
  Other Names: TECENTRIQ
  Arms: Dose Escalation Arm 1: Combination with atezolizumab Cohort 1; Dose Escalation Arm 1: Combination with atezolizumab Cohort 2; Dose Escalation Arm 1: Combination with atezolizumab Cohort 3; Dose Escalation Arm 2: Combination with atezolizumab and chemotherapy Cohort 1; Dose Escalation Arm 2: Combination with atezolizumab and chemotherapy Cohort 2; Dose Escalation Arm 2: Combination with atezolizumab and chemotherapy Cohort 3; Dose Expansion Arm 1: Combination with atezolizumab; Dose Expansion Arm 2: Combination with atezolizumab; Dose Expansion Arm 3: Combination with atezolizumab and chemotherapy
Drug: Standard of care chemotherapy — Chemotherapy to be administered according to the prescribing information.
  Arms: Dose Escalation Arm 2: Combination with atezolizumab and chemotherapy Cohort 1; Dose Escalation Arm 2: Combination with atezolizumab and chemotherapy Cohort 2; Dose Escalation Arm 2: Combination with atezolizumab and chemotherapy Cohort 3; Dose Expansion Arm 3: Combination with atezolizumab and chemotherapy

SUMMARY:
An Open Label, Multi-Center, Dose Escalation/Expansion, Phase 1/1b Study of IMU 201 (PD1-Vaxx), a B-Cell Immunotherapy as monotherapy or in combination with atezolizumab with or without chemotherapy, in Adults with Non-Small Cell Lung Cancer (IMPrinter).

DETAILED DESCRIPTION:
Investigational Medicinal Product, IMU-201, consists of drug substance, APi2568, which is a B-cell epitope (amino acids 92-110 from PD-1) linked to a promiscuous T-cell epitope (amino acid residues 288-302 from measles virus fusion protein) via a 4-amino acid linker (Gly-Pro-Ser-Leu), and combined with Water for Injection (WFI) forms the drug product, IMU-201, which becomes PD1-Vaxx when emulsified with excipient Montanide ISA 720 VG.

It is hypothesized that a polyclonal induced B-cell antibody response will be more effective or as effective with improved safety over current monoclonal antibody therapy.

This phase 1/1b study is an open-label dose escalation/dose expansion study designed to assess the safety, tolerability, immunogenicity and efficacy of IMU-201 (PD1-Vaxx). Phase 1 monotherapy dose-escalation of IMU-201 (PD1-Vaxx), will enroll approximately 9-18 patients and establish the optimal monotherapy biological dose (mBOD). Once established, the dose cohort will be expanded to enroll additional 10 patients at the mBOD dose level. Phase 1b, a combination dose-escalation of IMU-201 (PD1-Vaxx) with atezolizumab and with or without chemotherapy, will enroll approximately 18-36 patients and establish the optimal combotherapy biological dose (cBOD). Once established, the dose cohort will be expanded to enroll additional 30 patients at the cBOD dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years with histologically confirmed non-small-cell lung cancer (NSCLC) tumor stage IIIb not eligible for definitive treatment or stage IV
2. Prior treatment criterion for Monotherapy dose escalation and expansion: progressed on/after prior PD-1/PD-L1 containing regimen
3. Prior treatment criteria for Combination dose escalation arms:

   1. IMU-201 + atezolizumab, patients naïve to prior treatment or progressed on/after prior PD-1/PD-L1 containing regimen
   2. IMU-201 + atezolizumab + chemotherapy, patient naïve to prior treatment naive
4. Prior treatment criteria for Combination dose expansion arms:

   1. IMU-201 + atezolizumab, progressed on/after prior PD-1/PD-L1 containing regimen
   2. IMU-201 + atezolizumab, patients naïve to prior treatment
   3. IMU-201 + atezolizumab + chemotherapy, patients naïve to prior treatment
5. PD-L1 expression criteria (testing by 22C3, SP142, or SP263) for Monotherapy dose escalation and expansion: TPS/TC ≥ 50% or IC ≥ 10%. Patients with PD-L1 TPS/TC<50% or IC<10% expression may be included with agreement of Sponsor
6. PD-L1 expression criteria for Combination dose escalation arms:

   1. IMU-201 + atezolizumab, TPS/TC ≥ 50% or IC ≥ 10%
   2. IMU-201 + atezolizumab + chemotherapy, independent of PD-L1 expression
7. PD-L1 expression criteria for Combination dose expansion arms:

   1. IMU-201 + atezolizumab, TPS/TC ≥ 50% or IC ≥ 10%
   2. IMU-201 + atezolizumab, TPS/TC ≥ 50% or IC ≥ 10%
   3. IMU-201 + atezolizumab + chemotherapy, independent of PD-L1 expression
8. Life expectancy of at least 12 weeks in the opinion of the Investigator
9. Zubrod/ECOG score performance status 0-1
10. At least one measurable lesion as defined by RECIST 1.1 criteria.
11. Adequate hematologic, liver, and renal function

Exclusion Criteria:

1. Prior therapy for advanced NSCLC within 3 weeks prior to Day 1;
2. Continuous systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 2 weeks prior to first dose of study treatment.;
3. Any previous grade 3 or higher toxicity to a PD-1 inhibitor or PD-L1 inhibitor;
4. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required treatment with immunosuppressive agents or has current pneumonitis/interstitial lung disease;
5. Known brain metastases requiring steroid treatment, or signs and symptoms indicating suspected brain metastases;
6. Current or previous history of auto-immune disease;
7. NSCLC expressing epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), B-Raf proto-oncogene (BRAF) or ROS proto-oncogene 1 (ROS1) mutations who have not received appropriate therapies targeting these mutations and progress (if treatments are not available, patients who have NOT received appropriate therapies may be enrolled);
8. Prior organ transplant;
9. Concurrent active malignancy except for adequately controlled limited basal cell carcinoma of the skin;
10. History of uncontrolled seizures, central nervous disorders, or psychiatric disability judged by the Investigator to be clinically significant and precluding informed consent, participation in the study, or adversely affecting compliance to study drugs;
11. Active infection requiring intravenous antibiotics;
12. Known history of human immunodeficiency virus (HIV) infection or Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV Ribonucleic acid (RNA) [qualitative] is detected) infection;
13. Major surgery within 4 weeks prior to study entry. Minor surgery (excluding diagnostic biopsy) within 1 week prior to study entry;
14. Any vaccination within 2 weeks prior to starting study treatment;
15. Treatment with any investigational drug or participation in another investigational study within 3 weeks prior to first IMU-201 dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of IMU-201 graded per terminology criteria for adverse events (CTCAE) version 5.00 (Dose Escalation) | Baseline to Day 29
  Safety and Tolerability Measures include: Frequency of adverse events (AEs) graded per terminology criteria for adverse events (CTCAE) version 5.00.
Identify Optimal Biological Dose (OBD) with safety/tolerability graded per terminology criteria for adverse events (CTCAE) version 5.00 and Immuogenicity (Dose Escalation). | Baseline to Day 43
  Safety and Tolerability Measures: Adverse events (AEs); dose-limiting toxicities (DLTs) graded per terminology criteria for adverse events (CTCAE) version 5.00. Immunogenicity data for IMU-201 includes PD-1 specific antibody (IgG) titers.
Overall response rate (ORR) (Dose Expansion) | Baseline to documented progressive disease (Approximately 15 months)
  Efficacy of IMU-201 will be evaluated by overall response rate at OBD of IMU-201 measured as the proportion of participants with a best overall response of complete or partial response.

SECONDARY OUTCOMES:
Overall response rate (ORR) (Dose Escalation) | Baseline to documented progressive disease (Approximately 15 Months)
  Efficacy of IMU-201 will be evaluated by overall response rate at OBD of IMU-201 measured as the proportion of participants with a best overall response of complete or partial response.
Progression free survival (PFS) (Dose Escalation/Expansion) | Baseline to documented progressive disease or death due to any cause (Approximately 15 Months)
  Efficacy of IMU-201 will be evaluated by progression free survival at OBD of IMU-201.
Overall survival (OS) (Dose Escalation/Expansion) | Baseline to death from any cause (Approximately 15 Months)
  Efficacy of IMU-201 will be evaluated by overall survival at OBD of IMU-201.
Duration of response (DOR) (Dose Escalation/Expansion) | From date of earliest CR or PR until the date of first documented progression or death from any cause (Approximately 15 Months)
  Efficacy of IMU-201 will be evaluated by duration of response at OBD of IMU-201.

OTHER OUTCOMES:
Exploratory Outcome: Humoral immunogenicity of IMU-201 (Dose Escalation/Expansion) | Baseline to documented progressive disease (Approximately 15 Months)
  Humoral immunogenicity evaluated by PD-1 specific antibodies (IgG, IgM).
Exploratory Outcome: Cellular immunogenicity of IMU-201 (Dose Escalation/Expansion) | Baseline to documented progressive disease (Approximately 15 Months)
  Cellular immunogenicity evaluated by vaccine-specific cytokine levels as well as analysis of regulatory and effector T and B cells.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Ohio State University Medical Center, Columbus, Ohio
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Macquarie University, Macquarie, New South Wales
  - Cabrini Malvern Hospital, Melbourne, Victoria

REFERENCES:
- See also: Imugene Limited — https://www.imugene.com/